CLINICAL TRIAL: NCT03517748
Title: Evaluation of the Efficacy and Safety of DM05 Versus Optive™ on the Treatment of Moderate to Severe Ocular Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15E1122; 2016-A01843-48 (Other: ANSM)
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Because the comparator will be in commercial packaging, the blinding of the subject is not possible.
  However, the study will be blinded for the investigator: evaluations will be done by an independent investigator, different than the person who will distribute the product. Subjects will be identified by a patient number. Each patient number will be associated to a treatment number, according to a randomization list provided before the beginning of the clinical investigation, and randomized either in one of both treatment groups (DM05 or Optive®).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the investigational device: DM05 (Experimental): DM05 eye drops, multidose sterile emulsion, will be administered in the DM05 Arm at one to two drops instilled in each eye from 4 to 6 times per day during 84 days
  Interventions: Device: DM05 eye drops
- The comparative device : Optive™ (Active Comparator): Optive™ eye drops, multidose sterile solution, will be administered in the Optive Arm at one to two drops instilled in each eye from 4 to 6 times per day during 84 days
  Interventions: Device: Optive™ eye drops

INTERVENTIONS:
Device: DM05 eye drops — Ophthalmic use. One to two drops instilled in each eye from 4 to 6 times per day during 84 days of treatment.
  Arms: the investigational device: DM05
Device: Optive™ eye drops — Ophthalmic use. One to two drops instilled in each eye from 4 to 6 times per day during 84 days of treatment.
  Arms: The comparative device : Optive™

SUMMARY:
This study is a multicentric, comparative, randomized, investigator-blinded, in parallel groups study to demonstrate the non-inferiority of DM05 in comparison with Optive™, in terms of cornea and conjunctiva staining (Oxford score) on patients with moderate to severe ocular dryness, after 35 days of treatment.

DETAILED DESCRIPTION:
Evaluation of the non-inferiority of DM05 in comparison with OptiveTM, in terms of cornea and conjunctiva staining (Oxford score), on worse eye, between D0 and D35.

* Comparison of D35 versus D0 and D84 versus D0 for each product and comparison between products for the following parameters:

  * Evolution of cornea and conjunctiva staining (Oxford score) on worse eye.
  * Evolution of OSDI score (Ocular Surface Disease Index).
  * Evolution of Van Bijsterveld score (Lissamine green staining) in worse eye.
  * Evolution of Schirmer test result in worse eye.
  * Evolution of Tear film Break-Up Time (TBUT) in worse eye.
  * Evolution of ocular dryness severity by evaluation of each main symptom by the patient and total score of all symptoms
  * Evaluation of treatment performance by the investigator and the patient.
* Evaluation of the average frequency of use during 84 days for DM05 and OptiveTM.

Selection visit: D-14 to D-7

Wash-out period: 1 to 2 weeks with preservative-free 0.9% NaCl at 3 drops per day (Hydrabak®):

D0 : inclusion visit Follow-up visits: D35, D84

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female.
* Age: more than 18 years.
* Subject with a dry eye syndrome needing artificial tears in the 3 months preceding the inclusion.
* Subject having used only artificial tears without preservative (NaCl 0.9%, Hydrabak®) during 1 or 2 weeks before inclusion (at 3 drops per day).
* Diagnosis of moderate to severe ocular dryness defined by a score OSDI (Ocular Surface Disease Index) ≥18.
* Subject with at least one eye with:

  * Global ocular staining (cornea and conjunctiva) ≥4 and ≤9 (Oxford scale from 0 to 15)

AND one the following criteria:

* Schirmer test ≥ 3mm/5 min and ≤9mm/ 5 min OR
* Sum of 3 measurements of Tear film Break-Up Time (TBUT) ≤ 30s.

  * Subject, having given freely and expressly his/her informed consent.
  * Subject who is able to comply with the study requirements, as defined in the present protocol, at the Investigator's appreciation.
  * In France: subject being affiliated to a health social security system.
  * Female subjects of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject deprived of freedom by administrative or legal decision.
* Subject in a social or sanitary establishment.
* Major subject who is under guardianship or who is not able to express his consent.
* Subject being in an exclusion period for a previous study.
* Subject suspected to be non-compliant according to the Investigator's judgment.
* Subject wearing contact lenses during the study.
* Far best corrected visual acuity < 1/10
* Subject with severe ocular dryness with one of these conditions:

  * Eyelid or blinking malfunction
  * Corneal disorders not related to dry eye syndrome
  * Ocular metaplasia
  * Filamentous keratitis
  * Corneal neovascularization
* Subject with severe meibomian gland dysfunction (MGD)
* Within the last 3 months prior to the inclusion, history of ocular trauma, infection or inflammation not related to dry eye syndrome.
* Within the last 12 months, history of ocular allergy or ocular herpes.
* Refractive or cataract surgery within the last 6 months.
* Any laser other than refractive surgery within the last 3 months.
* Any troubles of the ocular surface not related to dry eye syndrome.
* Ocular hypertension or glaucoma needing an hypotonic treatment
* Subject having used artificial tears in the 6 hours preceding the inclusion visit.
* Use during the month preceding the inclusion or during the study of: isotretinoïd, cyclosporine, tacrolimus, sirolimus, pimecrolimus, punctual plugs.
* Any not stabilized systemic treatment, which can have an effect on performance or safety criteria, at the investigator appreciation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Demonstrate the non-inferiority of DM05 in comparison with OptiveTM, in terms of cornea and conjunctiva staining (Oxford score) on patients with moderate to severe ocular dryness, after 35 days of treatment. | 35 days
  Assess the ocular surface fluorescein staining score- mean change from Baseline in the study at D35 in ocular surface fluorescein stainig score according to a scale from zero to 15

SECONDARY OUTCOMES:
To assess the total ocular surface fluorescein staining score at D84 | 0 and 84 days
  Mean change from Baseline (D0) in the study eye and D84 in the total ocular surface fluoresceine staining score
Evolution of DEQ-5 score | 35 days
  Evolution from Baseline of DEQ-5 questionnaire scores at day 35
Evolution of DEQ-5 score | 84 days
  Evolution from Baseline of DEQ-5 questionnaire scores at day 84
Evolution of Van Bijterveld score ( lissamine green staining) | 35 Days
  Mean change from Baseline ( D0) and D 35 in the total Van Bijterveld score
Evolution of Van Bijterveld score ( lissamine green staining) | 84 days
  Mean change from Baseline ( D0) and D 84 in the total Van Bijterveld score
Volume tear fluid secretion as assessed by schirmer test | 35 days
  Mean change from Baseline ( D0) in Volume tear fluid secretion as assessed by schirmer test, at day 35
Volume tear fluid secretion as assessed by schirmer test | 84 days
  Mean change from Baseline ( D0) in Volume tear fluid secretion as assessed by schirmer test, at day 84
Evolution of Tear film Break-Up Time | 35 days
  Mean change from Baseline (D0) in the study eye in TFBUT at Day 35
Evolution of Tear film Break-Up Time | 84 days
  Mean change from Baseline (D0) in the study eye in TFBUT at Day 84
Global sum score of dry eye symptoms at visit 3 - mean change from Baseline at visit 3 ( D35) | 35 days
  Mean change from Baseline in the global sum score of dry eye symptoms at D35 : discomfort,burning, stinging,eye dryness sensation, itching,foreign body sensation,photophobia, blurred vision.Each graded from 0 to 10
Global sum score of dry eye symptoms at visit 4 - mean change from Baseline at visit 3 ( D84) | 84 days
  Mean change from Baseline in the global sum score of dry eye symptoms at D84 : discomfort,burning, stinging,eye dryness sensation, itching,foreign body sensation,photophobia, blurred vision.Each graded from 0 to 10
Global treatment performance score assessed by the investigator at visit 3 | 35 days
  Total Treatment performance score graded from 0 to 4
Global treatment performance score assessed by the investigator at visit 4 | 84 days
  Total Treatment performance score graded from 0 to 4
Global treatment performance score assessed by the patient at visit 3 | 35 days
  Total Treatment performance score graded from 0 to 4
Global treatment performance score assessed by the patient at visit 4 | 84 days
  Total Treatment performance score graded from 0 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baudouin, Pr, Principal Investigator — Hopital d Ophtalmologie des Quinze-vingts

IPD SHARING:
Plan to Share IPD: Undecided
Depending on any journal publication of the results

DOCUMENTS (2):
  • Study Protocol (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03517748/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03517748/SAP_001.pdf